CLINICAL TRIAL: NCT04601454
Title: DTM (TM) Low Energy Spinal Cord Stimulation (SCS) Study
Brief Title: DTM (TM) Spinal Cord Stimulation (SCS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20042
Record Dates: First submitted 2020-10-05; First posted 2020-10-23 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): Enrolled subjects are implanted with a rechargeable spinal cord stimulation system that is activated and programmed to on-label parameters.
  Interventions: Device: Spinal Cord Stimulation System

INTERVENTIONS:
Device: Spinal Cord Stimulation System — Rechargeable Implanted neurostimulation system (neurostimulator and leads) with on-label stimulation parameters.
  Other Names: Medtronic Intellis AdaptiveStim Neurostimulation System

SUMMARY:
Prospective, multi-center, open-label, post-market study to evaluate the efficacy and energy use of a low energy DTM™ (DTM-LE) SCS therapy for pain relief.

DETAILED DESCRIPTION:
This post market study will measure the following:

* Visual Analog Scale
* Programming Parameters

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to provide signed and dated informed consent
* Capable of comprehending and consenting in English
* Candidate per labeling for an SCS system as an aid in the management of chronic, intractable pain of the trunk and/or limbs
* Has moderate to severe back and leg pain
* Stable pain medications for back and leg pain for at least 28 days prior to enrollment
* Willing and able to comply with all study procedures and visits
* Willing and able to not increase their pain medications through the 3-Month visit
* Able to differentiate between pain associated with the indication for SCS implant and other types of pain

Exclusion Criteria:

* Previously trialed or implanted with a stimulator or intrathecal drug delivery system
* Expected to be inaccessible for follow-up
* Current diagnosis of moderate to severe central lumbar spinal stenosis with symptomatic neurogenic claudication
* Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results
* If female, is pregnant or is of child-bearing potential and unwilling to use a medically acceptable form of birth control during the study
* Has untreated major psychiatric comorbidity
* Serious drug-related behavioral issues
* Unable to achieve supine or prone position
* Classified as vulnerable or requires a legally authorized representative (LAR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Restorative Therapies Group Restorative Therapies Group, Study Director — Medtronic
Locations (13):
- United States (13):
  - IPM Medical Group, Walnut Creek, California
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Drez One LLC, Somerset, Kentucky
  - Carolinas Pain Center, Huntersville, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Oklahoma Pain Physicians, Oklahoma City, Oklahoma
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - Delaware Valley Pain and Spine Institute, Trevose, Pennsylvania
  - The Woodlands Pain Institute, Conroe, Texas
  - The Burkhart Research Institute for Orthopaedics, San Antonio, Texas
  - Sprintz Center for Pain, Shenandoah, Texas
  - Precision Spine Care, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation: Enrolled subjects are implanted with a rechargeable spinal cord stimulation system that is activated and programmed to on-label parameters.
  Spinal Cord Stimulation System: Implanted rechargeable neurostimulation system (neurostimulator and leads) with on-label stimulation parameters.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 57 (Total subjects)
Completed Per Protocol at the 12 Month Visit | 27 (Programmed to Differential Target Multiplex - Low Energy (DTM-LE) per protocol through the 12 month visit (secondary objective))
Completed | 32 (Programmed to Differential Target Multiplex - Low Energy (DTM-LE) per protocol through the 3 month visit (primary objective))
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: To characterize changes in overall (back and leg) pain intensity. Pain will be assessed using a VAS (0-10 cm) with 0 cm meaning "no pain" and 10 cm meaning "worst pain imaginable". Overall pain is defined as a combination of back and leg pain, but not pain from other body parts. Subjects will be asked to report their average pain intensity that is related to their SCS device treatment "in the last 24 hours" by marking a line perpendicular to the VAS line at the point that represents their pain intensity.
Time Frame: Baseline to 3 Months
Measure: Mean (Standard Deviation); unit: Centimeter
Groups:
- Spinal Cord Stimulation: Enrolled subjects are implanted with a rechargeable spinal cord stimulation system that is activated and programmed to on-label parameters.
  Spinal Cord Stimulation System: Implanted rechargeable neurostimulation system (neurostimulator and leads) with on-label stimulation parameters per protocol. Outcome measures were provided at baseline and 3 month visits and compared. Difference in VAS was calculated such that a negative value indicates a reduction in pain related to the VAS from baseline.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 32
Centimeter | -3.9 (2.45)

2. Secondary Outcome: Programming Parameters: Frequency in Hertz (Hz)
Description: To characterize programming parameters associated with energy use. Subject's programmed frequency settings will be summarized using the minimum and maximum frequency across all subjects. Programming methodology for this study included up to four active program frequencies for each subject.
Time Frame: 12 Month
Population: Frequencies reported represent the range of the sum of active programs across all subjects. Patients analyzed included those who completed the study per protocol at the 12 month visit.
Measure: Number; unit: Hertz (Hz)
Groups:
- Spinal Cord Stimulation: Enrolled subjects are implanted with a rechargeable spinal cord stimulation system that is activated and programmed to on-label parameters.
  Spinal Cord Stimulation System: Implanted rechargeable neurostimulation system (neurostimulator and leads) with on-label stimulation parameters per protocol.
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 27
Hertz (Hz)
  Range Minimum | 250.0
  Range Maximum | 300.0

3. Secondary Outcome: Programming Parameters: Pulse Width in Microseconds (µs)
Description: To characterize programming parameters associated with energy use. Subject's programmed Pulse Width settings will be summarized using the minimum and maximum Pulse Width across all subjects. Programming methodology for this study included up to four active program frequencies for each subject.
Time Frame: 12 Month
Population: Pulse Width in microseconds (µs) reported represent the range of active programs across all subjects. Patients analyzed included those who completed the study per protocol at the 12 month visit.
Measure: Number; unit: microseconds (µs)
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 27
microseconds (µs)
  Range Minimum | 200.0
  Range Maximum | 200.0

4. Secondary Outcome: Programming Parameters: Amplitude (Intensity) in Milliamp (mA)
Description: To characterize programming parameters associated with energy use. Subject's programmed Amplitude settings will be summarized using the minimum and maximum Amplitude across all subjects. Programming methodology for this study included up to four active program frequencies for each subject.
Time Frame: 12 Month
Population: Amplitude (intensity) in milliamp (mA) reported represent the range of active programs across all subjects. Patients analyzed included those who completed the study per protocol at the 12 month visit.
Measure: Number; unit: milliamp (mA)
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 27
milliamp (mA)
  Range Minimum | 0.70
  Range Maximum | 7.3

5. Secondary Outcome: Programming Parameters: Impedance Range in Ohms
Description: To characterize programming parameters associated with energy use. Subject's programmed Impedance settings will be summarized using the minimum and maximum Impedance across all subjects. Programming methodology for this study included up to four active program frequencies for each subject.
Time Frame: 12 Month
Population: Impedance (ohms) reported represent the range of active programs across all subjects. Patients analyzed included those who completed the study per protocol at the 12 month visit.
Measure: Number; unit: ohms
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 27
ohms
  Range Minimum | 670.0
  Range Maximum | 2,020.0

ADVERSE EVENTS:
Time Frame: Adverse events will be collected throughout the study duration, starting at the time of signing the informed consent through the subjects12 month visit, or study completion.
Description: All device-related, procedure-related, and therapy-related adverse events will be considered reportable for this study. Adverse events will be collected on an Adverse Event Case Report Form.
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 12/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Cord Stimulation (N=57)
Implant site infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Cord Stimulation (N=57)
Medical device site oedema (General disorders) | 1
Medical device site pain (General disorders) | 2
Incision site complication (Injury, poisoning and procedural complications) | 1
Incision site swelling (Injury, poisoning and procedural complications) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Lead dislodgement (Product Issues) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT04601454/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04601454/SAP_003.pdf